CLINICAL TRIAL: NCT01136876
Title: Pilot Study to Evaluate Kidney Damage Measured by Neutrophil Gelatinase-Associated Lipocalin as New Biomarker in Patients With Moderate Fall in eGFR Undergoing Percutaneous Coronary Intervention With IOPAMIDOL Injection 370 or IODIXANOL 320
Brief Title: Kidney Damage in Patients With Moderate Fall in eGFR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: IOP-117
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Results first posted 2013-12-30 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2013-09

CONDITIONS: Coronary Artery Stenosis
MeSH Terms: conditions — Coronary Stenosis | interventions — Iopamidol; iodixanol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Iopamidol (Active Comparator): Non-ionic low-osmolar iodinated contrast media
  Interventions: Drug: Iopamidol
- Iodixanol (Active Comparator): Non-ionic iso-osmolar iodinated contrast media comparator
  Interventions: Drug: Iodixanol-320

INTERVENTIONS:
Drug: Iopamidol — Iopamidol 370, one time administration for percutaneous coronary intervention
  Other Names: Isovue-370
  Arms: Iopamidol
Drug: Iodixanol-320 — Iodixanol-320 single administration for percutaneous coronary intervention procedure
  Other Names: Visipaque 320
  Arms: Iodixanol

SUMMARY:
To compare Iopamidol injection 370 and Iodixanol 320 in evaluating Neutrophil Gelatinase-Associated Lipocalin (NGAL) in patients with moderate fall in eGFR

DETAILED DESCRIPTION:
This is a pilot study having a randomized, double-blind parallel group comparison of two iodinated contrast agents used during percutaneous coronary intervention (PCI). All patients enrolled must have eGFR greater than or equal to 30 mL/min and less than or equal to 59 mL/min. Statistical summaries will be presented to analyze the various lab tests results for the two groups.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age and provides informed consent
* Scheduled to undergo percutaneous coronary intervention
* Documented pre-dose Estimated glomerular filtration rate (eGFR) of greater than or equal to 30 mL/min/1.73 m squared and less than or equal to 59 mL/min/1.73 m squared

Exclusion Criteria:

* Pregnant or lactating females
* Severe congestive heart failure
* History of hyperthyroidism;
* Unstable renal function
* Emergency PCI
* History of hypersensitivity to iodinated contrast agents
* Receiving diuretics to prevent acute renal injury

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Luigia Storto, MD, Study Director — Bracco Diagnostics, Inc
Locations (4):
- United States (3):
  - Research Cooperative, St. John's Hospital, Springfield, Illinois
  - UMDNJ - RWJ Medical School, New Brunswick, New Jersey
  - The Institute for Clinical Research at Holy Name Medical Center, Teaneck, New Jersey
- Montreal Heart Institute, Montreal, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Iodixanol 320: Iodixanol 320, a non-ionic iso-osmolar iodinated contrast media comparator, was administered as a single 652 mg dose for percutaneous coronary intervention procedure
- Iopamidol 370: Iopamidol 370, a non-ionic low-osmolar iodinated contrast media, was administered as a single 755 mg dose for percutaneous coronary intervention procedure
Period: Overall Study
Arm/Group | Iodixanol 320 | Iopamidol 370
Started | 28 | 29
Completed | 23 | 18
Not Completed | 5 | 11
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 3 | 5
Not completed — Missing NGAL measurement | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Iodixanol 320: Iodixanol 320 Non-ionic iso-osmolar iodinated contrast media comparator: single administration for percutaneous coronary intervention procedure
- Iopamidol 370: Iopamidol 370 Non-ionic low-osmolar iodinated contrast media: single administration for percutaneous coronary intervention procedure
- Total: Total of all reporting groups
Arm/Group | Iodixanol 320 | Iopamidol 370 | Total
Number analyzed (Participants) | 28 | 29 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (7.4) | 73.3 (10.0) | 72.2 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 19 | 17 | 36
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 38
  Canada | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Impact on the Trajectory of Serum and Urinary Neutrophil Gelatinase-associated Lipocalin (NGAL) Following Administration
Description: Mean change from baseline values for serum NGAL at 2,4,6,24,48, and 72 hours, and urine NGAL at 2,4,6,24, and 48 hours following the administration of contrast media.
Time Frame: Baseline and 2, 4, 6, 24, 48,and 72 hours post-dose
Population: A total of 41 patients met the evaluable criteria for NGAL analysis, 18 patients that were administered iopamidol 370, and 23 patients that were administered iodixanol 320.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Iodixanol 320 Serum NGAL: Serum NGAL (ng/mL) mean change from baseline at 2,4,6,24,48, and 72 hours post-administration of iodixanol 320
- Iodixanol 320 Urine NGAL: Urine NGAL (ng/mL) mean change from baseline at 2,4,6,24, and 48 hours post-administration of iodixanol 320
- Iopamidol 370 Serum NGAL: Serum NGAL (ng/mL) mean change from baseline at 2,4,6,24,48, and 72 hours post-administration of iopamidol 370
- Iopamidol 370 Urine NGAL: Urine NGAL (ng/mL) mean change from baseline at 2,4,6,24,and 48 hours post-administration of iopamidol 370
Arm/Group | Iodixanol 320 Serum NGAL | Iodixanol 320 Urine NGAL | Iopamidol 370 Serum NGAL | Iopamidol 370 Urine NGAL
Number analyzed (Participants) | 23 | 23 | 18 | 18
ng/mL
  2 hours post-dose | -27.76 (51.89) | -11.11 (16.32) | -11.84 (30.49) | -8.23 (9.90)
  4 hours post-dose | -27.06 (46.03) | -10.68 (15.10) | -14.66 (42.24) | -4.87 (15.06)
  6 hours post-dose | -15.83 (47.06) | -6.88 (10.61) | -17.61 (37.28) | -7.70 (7.44)
  24 hours post-dose | 15.89 (78.14) | -5.85 (15.68) | 35.06 (85.39) | 4.46 (18.03)
  48 hours post-dose | 22.88 (59.34) | -0.85 (16.57) | 54.54 (52.62) | 11.18 (21.60)
  72 hours post-dose | 22.32 (60.51) | NA (NA) — Urine NGAL not measured at 72 hours post-dose as per protocol. | 33.18 (52.92) | NA (NA) — Urine NGAL not measured at 72 hours post-dose as per protocol.

ADVERSE EVENTS:
Time Frame: All adverse events that occurred from the time the patient signed the Informed Consent Form through 2 hours post dose were recorded.
Groups:
- Iopamidol 370: Iopamidol 370 Non-ionic low osmolar iodinated contrast media: single administration for percutaneous coronary intervention
Arm/Group | Iodixanol 320 | Iopamidol 370
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/29
Other Adverse Events (participants affected / at risk) | 0/28 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days